CLINICAL TRIAL: NCT01575860
Title: Maintenance Lenalidomide Therapy After Autologous Stem Cell Transplant in Patients With High Risk Relapsed/Refractory Lymphomas
Brief Title: Maintenance Lenalidomide in Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 11411
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma
Keywords: biopsy-proven diagnosis; completed at least 2 cycles of salvage chemotherapy; showing PET positive residual lesions
MeSH Terms: conditions — Lymphoma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I/II (Maintenance Lenalidomide in Lymphoma) (Experimental): Total of 24 cycles of lenalidomide. Subjects received a starting daily dose of 10mg lenalidomide on days 1 through 28 of each 28 day cycle. Subjects initiated lenalidomide 28-100 days post-ASCT.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide, 10mg, oral tablets, daily
  Other Names: Revlimid, CC-5013

SUMMARY:
This study is being conducted to evaluate the overall safety of lenalidomide (also known as Revlimid) in patients with lymphoma, and to determine whether it is effective in preventing this disease from returning after stem cell transplant. This study will also determine the dose of lenalidomide that can be given without causing severe side effects. Lenalidomide has not been approved by the U.S. Food and Drug Administration (FDA) for the treatment of lymphoma. At least 28 people will be enrolled on this study at the University of Pennsylvania.

DETAILED DESCRIPTION:
Describe succinctly and clearly the past findings which justify the plan for this project. A summary of the relevant literature in the area of interest and reports of previous studies should be included.

For majority of lymphoma patients who relapse after complete response or who are primary refractory to initial treatment, a combination of salvage chemotherapy followed by high dose chemotherapy and ASCT is considered the standard of care. Sensitivity to salvage chemotherapy affects the outcome after ASCT. Traditionally, the response to salvage chemotherapy prior ASCT was determined by conventional computed tomography (CT) scans using size criteria. In the past several years, it has been shown that functional imaging with PET scans using fluorodeoxyglucose (FDG) provides additional information to anatomic imaging with CTs. Recently, PET scans have been incorporated into the response assessment as published by the Imaging Subcommittee of International Harmonization Project in Lymphoma. These days, most institutions use PET/CT scans which incorporate functional imaging with PET scan fused with low dose non-contrast enhanced CT scan.

We have previously reported the outcome of patients with relapsed/refractory lymphomas who continued to have residual FDG avid PET (positive) lesions after salvage chemotherapy and prior to ASCT. This group of patients included those who had excellent anatomic response by size criteria, but continued to have persistent hypermetabolic FDG activity within the residual lesions. We found that PET positive patients have an extremely poor chance of durable remission after ASCT. In the PET negative group, the median PFS was 19 months with 54% of patients without progression at 12 months after ASCT. In the PET positive group, the median PFS was 5 months with only 7% of patients without progression at 12 months after ASCT. We concluded that, for patients with PET positive residual disease after salvage chemotherapy and prior to ASCT, novel therapeutic approaches and agents need to be investigated.

Lenalidomide is a proprietary IMiD® compound of Celgene Corporation. IMiD® compounds have both immunomodulatory and anti-angiogenic properties which could confer antitumor and antimetastatic effects. Although the exact antitumor mechanism of action of lenalidomide is unknown, a number of mechanisms are postulated to be responsible for lenalidomides activity against hematological malignancies. Lenalidomide has been demonstrated to possess anti-angiogenic activity through inhibition of bFGF, VEGF and TNF-alpha induced endothelial cell migration, due at least in part to inhibition of Akt phosphorylation response to bFGF. In addition, lenalidomide has a variety of immunomodulatory effects. Lenalidomide stimulates T cell proliferation, and the production of IL-2, IL-10 and IFN-gamma, inhibits IL-1 beta and IL-6 and modulates IL-12 production. Up-regulation of T cell derived IL-2 production is achieved at least in part through increased AP-1 activity. The increased levels of circulating cytokines augment natural killer cell number and function, and enhance natural killer cell activity.

Clinical activity of lenalidomide in various lymphoma subtypes has been documented in several phase II trials. In patients with relapsed/refractory mantle cell lymphoma, the overall response rate (ORR) was 53% with PFS at 12 month 40%. In patients with aggressive lymphoma (mostly diffuse large B-cell subtype), the ORR was 35% with PFS at 12 months about 25%. There also have been many case reports of patients who achieved durable complete response to lenalidomide after failing multiple cytotoxic chemotherapy regimens.

Most clinical studies of lenalidomide in patients with active lymphoma used dose of 25 mg daily on days 1-21 in 28 day cycle which is the dosing recommended for active multiple myeloma. While lenalidomide was well tolerated in the lymphoma studies, the dose of 25 mg is associated with high risk of developing cytopenias including grade 3 neutropenia in 25-40% of patients and thrombocytopenia in 12-20%. Our group reported that low dose lenalidomide at 10 mg daily (continuous dosing) in combination with weekly dexamethasone can be effective in patients with active relapsed/refractory low grade and mantle cell lymphomas. The continuous dose of 10 mg daily has also been used in treatment of chronic lymphocytic leukemia/small lymphocytic lymphoma.

Lenalidomide has been used as maintenance therapy in multiple myeloma, but there is limited experience with maintenance lenalidomide in lymphoma patients. Two large clinical trials of maintenance lenalidomide in patients with multiple myeloma after ASCT have shown benefit in PFS over observation. These studies used daily dosing of lenalidomide at 10 mg or 15 mg which were well tolerated over long term administration.

Revlimid® (lenalidomide) is currently indicated for the treatment of patients with transfusion-dependent anemia due to Low- or Intermediate-1-risk myelodysplastic syndromes associated with a deletion 5q cytogenetic abnormality with or without additional cytogenetic abnormalities. Revlimid® is also approved in combination with dexamethasone for the treatment of patients with multiple myeloma that have received at least one prior therapy.

The most frequently reported adverse events reported during clinical studies with lenalidomide in oncologic and non-oncologic indications, regardless of presumed relationship to study medication include: anemia, neutropenia, thrombocytopenia and pancytopenia, abdominal pain, nausea, vomiting and diarrhea, dehydration, rash, itching, infections, sepsis, pneumonia, UTI, Upper respiratory infection, atrial fibrillation, congestive heart failure, myocardial infarction, chest pain, weakness, hypotension, hypercalcemia, hyperglycemia, back pain, bone pain, generalized pain, dizziness, mental status changes, syncope, renal failure, dyspnea, pleural effusion, pulmonary embolism, deep vein thrombosis, CVA, convulsions, dizziness, spinal cord compression, syncope, disease progression, death not specified and fractures.

Complete and updated adverse events are available in the Investigational Drug Brochure and the IND Safety Letters.

Rationale for Treatment in this Setting:

Our previously reported data and similar studies from other institutions indicate that patients with PET positive lesions after salvage chemotherapy and prior ASCT do very poorly. In our study, patients with residual PET positive lesions before ASCT had median PFS of 5 months with only 7% of patients without progression at 12 months after ASCT. It can be speculated that patients with PET positive lesions prior ASCT harbor chemotherapy resistant lymphoma cells in their tumors. Since the mechanism of action of lenalidomide differs from traditional cytotoxic chemotherapy, the use of this novel agent in this group of patients is an attractive concept. The immunomodulary properties of lenalidomide over the maintenance period of 24 months could improve the overall outcome of patients following ASCT. Since there is a valid concern that lenalidomide could cause severe cytopenias when used early after ASCT, we proposed to administer dose 10 mg of lenalidomide daily with an option of dose modification to 5 mg daily according to previously defined toxicity criteria. The daily maintenance dosing of lenalidomide at 10 mg has been used in patients with multiple myeloma after ASCT and improved PFS in two large randomized trials.

ELIGIBILITY:
Inclusion Criteria:

SCREENING STEP A:

1. Able to understand and voluntarily sign the informed consent form.
2. Aged greater or equal to 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Biopsy-proven diagnosis of lymphoma (including diffuse large B-cell, mantle cell, follicular, marginal zone, peripheral T cell, small lymphocytic lymphoma with large cell transformation, and Hodgkin lymphomas).
5. Completion of at least 2 cycles of salvage chemotherapy, with pre-ASCT PET/CT imaging showing PET positive residual lesion(s) (SUV greater than 2.5).
6. Disease free of other malignancies for greater or equal to 2 years with exception of basal cell and squamous cell carcinomas of the skin, or carcinoma in situ of the cervix or breast.

NOTE: Patients who successfully complete high dose-chemotherapy and ASCT will proceed to Screening Step B, provided that they achieve hematologic recovery within 100 days of ASCT (see below).

SCREENING STEP B (performed between days 28-100 post-ASCT):

1. Completion of high-dose chemotherapy with ASCT.
2. Hematologic recovery at 28-100 days after ASCT (defined as ANC greater or equal to 1,000 and platelet count greater or equal to 60,000).
3. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
4. ECOG performance status of less than or equal to 2 at study entry (see Appendix B).
5. Patients undergoing planned consolidative radiation therapy must be finished with the therapy by day 100 after ASCT.
6. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 to 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
7. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (warfarin or low molecular weight heparin may be used for patients intolerant of aspirin or at the discretion of the treating physician).

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females (lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of initiating treatment with lenalidomide.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum, a blistering or desquamating rash, while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or therapies during study treatment.
9. Known seropositive for or active viral infection with human immunodeficiency virus (HIV) or hepatitis B virus (HBV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2018-05-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Svoboda, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Jakub Svoboda, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Maintenance Lenalidomide in Lymphoma: Total of twenty-four (24) 28-day cycles of Lenalidomide, 10mg, oral tablets, daily
Period: Overall Study
Arm/Group | Maintenance Lenalidomide in Lymphoma
Started | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Progression Prior to Lenalidomide Maint. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Maintenance Lenalidomide in Lymphoma
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 51 [29 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Lymphoma sub-type [Count of Participants; unit: Participants]
  Hodgkin Lymphoma | 2
  Diffuse Large B-Cell, Activated B-Cell subtype | 1
  Diffuse Large B-Cell, Germinal Center subtype | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose-limiting Toxicities
Description: Dose-limiting toxicity (DLT) is defined as any grade 3 toxicity or higher that occurs during the first 28 days of therapy and is possibly, probably, or definitely related to lenalidomide maintenance.
Time Frame: 28 days (Cycle 1)
Population: Eight (8) participants were enrolled: one (1) participant withdrew consent prior to completing Cycle 1; one (1) participant progressed prior to initiating lenalidomide maintenance; a total of six (6) subjects were evaluated for dose-limiting toxicities.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Lenalidomide in Lymphoma
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) is defined as days from start of high dose chemotherapy to first documented progression of disease, death due to any cause or last patient contact.
Time Frame: 12 months from start of lenalidomide maintenance
Population: Eight (8) participants were enrolled: one (1) participant withdrew consent prior to completing Cycle 1; one (1) participant progressed prior to initiating lenalidomide maintenance; six (6) participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Lenalidomide in Lymphoma
Number analyzed (Participants) | 6
Participants
  Participants without Disease Progression | 4
  Participants with Disease Progression | 2

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as days from start of high dose chemotherapy to death due to any cause or last patient contact.
Time Frame: 12 months from the start of lenalidomide maintenance
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Lenalidomide in Lymphoma
Number analyzed (Participants) | 6
Participants
  Participants Alive | 4
  Participants Deceased | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from each subject's first dose of lenalidomide to twenty-eight days following each subject's last dose of lenalidomide, or upon resolution of any treatment-related adverse events, should their duration extend beyond the 28-day reporting period up to 28 days +/- 7 days after participant study discontinuation.
Groups:
- Maintenance Lenalidomide in Lymphoma: Total of twenty-four (24) 28-day cycles of lenalidomide, 10mg, oral tablets, daily
  Lenalidomide: Lenalidomide, 10mg, oral tablets, daily
Arm/Group | Maintenance Lenalidomide in Lymphoma
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Lenalidomide in Lymphoma (N=6)
Fatigue (Grade 1) (General disorders) | 1 (1)
Fatigue (Grade 2) (General disorders) | 1 (1)
Cough (Grade 2) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypogammaglobunemia (Immune system disorders) | 1 (1)
White blood cell decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
The sample size of Phase 1 of Maintenance Lenalidomide in Lymphoma is small. The results need to be confirmed in a larger group of subjects. The trial was prematurely terminated by the Sponsor due to poor accrual. Phase II was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT01575860/Prot_SAP_000.pdf